CLINICAL TRIAL: NCT04313725
Title: An Evaluation of Tangible Boost Replenishing System for Patients With Stevens Johnson Syndrome, Sjogren's Syndrome, and Graft Versus Host Disease
Brief Title: Evaluation of Tangible Boost for Patients With Stevens Johnson Syndrome, Sjogren's Syndrome, and Graft Vs Host Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow enrollment and difficulty getting patients to complete the study visits (significantly impacted by COVID-19 pandemic)
Sponsor: Tangible Science (Industry)
Collaborators: Boston Sight (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DOC-55
Record Dates: First submitted 2020-03-16; First posted 2020-03-18 (Actual); Last update posted 2025-09-16 (Actual); Status verified 2025-09

CONDITIONS: Stevens-Johnson Syndrome; Graft Versus Host Disease in Eye; Sjogren's Syndrome; Dry Eye
Keywords: contact lens care
MeSH Terms: conditions — Stevens-Johnson Syndrome; Sjogren's Syndrome; Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Test and placebo treatment kits will be randomized by the sponsor prior to sending to clinical site.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Boost (Experimental): Subjects will use the Tangible Boost treatment on their lenses monthly throughout the study.
  Interventions: Device: Tangible Boost
- Placebo (Placebo Comparator): Subjects will use a Placebo treatment (saline) on their lenses monthly throughout the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Device: Tangible Boost — Patients will perform a monthly Tangible Boost treatment on their Hydra-PEG treated contact lenses.
  Arms: Boost
Other: Placebo — Patients will perform a monthly placebo (saline) treatment on their Hydra-PEG treated contact lenses.
  Arms: Placebo

SUMMARY:
The goal of this research is to determine if the Tangible Boost system adequately replenishes the Hydra-PEG coating on the surface of a rigid contact lens.

Hydra-PEG is a coating for soft and rigid contact lens, primarily composed of polyethylene glycol-based hydrogel, which is covalently bound to the surface of a contact lens. The Hydra-PEG coating is intended to improve wettability and comfort with contact lenses and is currently FDA approved on a number of contact lenses. For patients with Stevens Johnson Syndrome (SJS) (SS), or Graft versus Host disease (GVHD), diminished efficacy of the Hydra-PEG coating can lead to significant decline in satisfaction with the lenses over time. This is a prospective study to evaluate the efficacy of Tangible Boost, a monthly conditioning solution, to replenish the Hydra-PEG coating on rigid gas permeable contact lenses for patients with SJS, GVHD, and SS. Outcomes from this patient population will be compared to patients with dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

* Written Informed Consent has been obtained prior to any study-related procedures taking place
* Written documentation has been obtained in accordance with the relevant county and local privacy requirements, where applicable
* Male or female
* 18 years of age and older prior to the initial visit
* Is a new or established wearer of PROSE lenses with optimized lens fit prior to enrollment in the study
* Has been diagnosed with Dry Eye Syndrome, SJS, SS, or GVHD
* In the opinion of the investigator, the subject has the ability to follow study instructions
* In the opinion of the investigator, the subject has the ability to complete all study procedures and visits

Exclusion Criteria:

* aphakic (i.e., missing their natural lens inside the eye)
* Is currently participating in any other type of eye-related clinical or research study
* Is pregnant or nursing as reported by the subject
* Has a condition or is in a situation which, in the investigator's opinion, may put the subject at significant risk, may confound study outcomes, or may significantly interfere with the subject's participation in the study.
* Has a known and self-reported allergy to the following substances: polyethylene glycol, polyvinyl alcohol, triethanolamine, polyquaternium-1, or edetate disodium, which are components of the Tangible Boost and Hydra-PEG systems or care regimen.
* Has had previous ocular surgery within the past 12 weeks
* Adults unable to consent (including adults unable to read and understand English)
* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Employees of BostonSight

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-02-24 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Visual Acuity | 3 months
  Snellan visual acuity
Visual Acuity | 6 months
  Snellan visual acuity
Contact Lens Comfort | 3 months
  OSDI plus additional specific questions
Contact Lens Comfort | 6 months
  OSDI plus additional specific questions
Ocular Surface Staining | 3 months
  Sodium fluorescein staining will be used to evaluate ocular surface damage indicated by cell damage or death. Corneal staining will be scored using the Oxford grading scale.
Ocular Surface Staining | 6 months
  Sodium fluorescein staining will be used to evaluate ocular surface damage indicated by cell damage or death. Corneal staining will be scored using the Oxford grading scale.
Tear break up time | 3 months
  Seconds required for tear film to begin to break up
Tear break up time | 6 months
  Seconds required for tear film to begin to break up

SECONDARY OUTCOMES:
Contact lens fit characteristics | 6 months
  Changes in apical clearance, limbal clearance, scleral landing evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Karen Carrasquillo, OD, PhD, Principal Investigator — Boston Sight
Locations (1):
- Boston Sight, Needham, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No